CLINICAL TRIAL: NCT06368271
Title: Acute Effects of Dietary Medium-chain Fatty Acids on Llipid Profile
Brief Title: Acute Effects of Dietary Medium-chain Fatty Acids on Lipid Profile
Acronym: Lipidomix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lipidomix
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Healthy Nutrition; Diet, Healthy
Keywords: medium-chain fatty acids; lipidomics; acute intervention

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blinded crossover design. Participants ingest Medium-chain-fatty acids (MCT) or Long-chain fatty acids (LCT) oil on two test days with one-week period between the experimental days. The day prior to the experimental days, the participants consume a eucaloric control diet, and abstain from alcohol and vigorous physical activity to ensure similar conditions on experimental days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intake of fatty acids (Experimental): ,Participants ingest a test drink containing 35g of MCT or LCT oil diluted in 100g of low-fat, low-carb cocoa milk) within five min. Blood and oxygen uptake are obtained frequently during the following 4 hours.
  Interventions: Dietary Supplement: Lipidomics

INTERVENTIONS:
Dietary Supplement: Lipidomics — Health beneficial effects of medium-chain fatty acids

SUMMARY:
In the present study the plasma lipid profile was elucidated in healthy, lean males by the use of lipidomic analysis in the hours after an acute intake of medium-chain fatty acids (MCT) and long chain fatty acids (LCT),, respectively. In addition oxygen uptake was measured to study energy turnover.

DETAILED DESCRIPTION:
Four participants ingested MCT or LCT oil on two test days with one-week period between the experimental days. The day prior to the experimental days, the participants consumed a eucaloric control diet, and abstained from alcohol and vigorous physical activity to ensure similar conditions on experimental days.

On the test days, participants arrived by passive transport in the overnight fasted state (12 h) at 8 a.m., and a catheter was inserted into an antecubital vein. Following 30 min in supine rest, an overnight-fasted, basal venous blood sample was obtained. Subsequently, participants ingested the same test drink as in study 1 (containing 35g of MCT or LCT oil diluted in 100g of low-fat, low-carbohydrate cocoa milk) within five min. 100 ml water was provided together with the test drink. Venous blood samples were drawn every 30 min for the first two hours and every 60 minutes for the last two hours following intake. Participants rested in a bed throughout the test day. this This process was repeated on the second test day.

ELIGIBILITY:
Inclusion Criteria:

healthy males BMI:20-27 recreationally physical active non-smoker no medicine

-

Exclusion Criteria:

* high habitual intake of MCT-rich foods as coconut, coconut oil and dairy products

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Meal test including medium-chain fatty acids | 0-4 hours
  In this study the effect of an acute intake of MCT oil compared with the intake of LCT (containing 35g of MCT or LCT oil diluted in 100g of low-fat, low-carb cocoa milk ) on the plasma lipid profile is studied in healthy men. Blood is obtained postprandially ( frequently during 4 hours) and analyzed for the plasma lipid profile

SECONDARY OUTCOMES:
Resting metabolic rate | 0-4 hours
  The secondary outcome of this study is to investigate the effect of an acute intake of MCT or LCT oil (35g of MCT or LCT) on resting metabolic rate in healthy lean men

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, D.sci, PhD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen
  - Department of Nutrition, Exercise and Sports, Copenhagen